CLINICAL TRIAL: NCT00865267
Title: A Single-blind, Single Exposure Study, to Evaluate the Vasoconstriction Activity of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects: Dose Ranging Study
Brief Title: The Dose-response Study of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Christine Winslow, Director of Clinical Development, Actavis Inc
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: DP03-685
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Vasoconstriction; Halobetasol; Healthy adult subjects
MeSH Terms: interventions — halobetasol; Ointments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Ultravate® 0.05% ointment, single exposure
  Interventions: Drug: Ultravate® 0.05% ointment, single exposure

INTERVENTIONS:
Drug: Ultravate® 0.05% ointment, single exposure — A: Experimental Subjects received Bristol-Myers Squibb Company formulated products
  Other Names: Halobetasol

SUMMARY:
The purpose of this study is to determine the duration of application of halobetasol propionate 0.05% ointment to be used in a definitive study of bioequivalence of to formulations of this ointment.

Part A: To validate vasoconstrictor assay precision.

Part B: To evaluate the dose response vasoconstriction profile of Ultravate® 0.05% ointment at different dose durations over a short period of time (0.17 - 4 hrs).

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: A single blind, single-exposure study on healthy adult male and female subjects.

Official Title: A Single-blind, Single Exposure Study, to Evaluate the Vasoconstriction Activity of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects: Dose Ranging Study

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Vasoconstrictor Response

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study, is willing to participate, and gives written informed consent.
* Subject demonstrates adequate vasoconstriction to the screening topical corticosteroid Halobetasol propionate 0.05% Ointment.
* Subject is a non-smoking (minimum of 14 days), male or female, ages of 18 - 65 years, inclusive.
* Subject is within 20% of their ideal body weight as defined by the 1999 Metropolitan Life Insurance Company Height and Weight Tables.
* Subject is judged by the Investigator to be healthy on the basis of pre-study medical history.
* Subjects of child-bearing potential agree to use an acceptable method of birth control during study participation (e.g. abstinence, any prescribed birth control method, double barrier method, Le. condom plus foam, condom plus diaphragm).
* Subject is willing to refrain from excessive consumption of sodium in food or beverage 48hrs before and for the duration of the study.
* Subject is willing to shower using the same soap/cleansers for the duration of the study.
* Subject is willing to follow study restrictions.

Exclusion Criteria:

* Subject has a past or current medical condition that might significantly affect pharmacodynamic response to topical corticosteroids.
* Subject has clinically significant hypertension or circulatory disease.
* Subject is taking any medication on a regular basis that could modulate blood flow (constrictor or dilator), with the exception of any prescribed birth control method and hormone replacement therapy. Examples of such drugs include nitroglycerin, anti-hypertensives, antihistamines, NSAIDs, aspirin, phenylpropanolamine, or phentolamine.
* Subject is planning to use any exclusionary over-the-counter (OTC) medications within 48 hours prior to or throughout the study that could modulate blood.
* Subject has a history of sensitivity/allergy to the ingredients found in the test formulations or has a history of adverse reactions to topical or systemic corticosteroids.
* Subject has a significant history of allergy to soaps, lotions, emollients, creams, ointments, cosmetics, adhesives, or latex.
* Subject has a history of significant skin conditions or disorders, for example, psoriasis, atopic dermatitis, actinic keratosis, etc.
* Subject has an obvious difference In skin color between arms or the presence of a skin condition, scar tissue, tattoo or coloration that would interfere with placement of test sites, their assessments or could compromise the safety of the subject.
* Subject has used topical medications on the ventral forearms within 1 month prior to dosing.
* Subject has used a tobacco product within 14 days of study conduct.
* Subject has a clinically significant history of drug abuse or alcoholism.
* Subject has donated or received blood within 30 days prior to dosing.
* Subject's caffeine intake is greater than 500 mg per day (1 cup of coffee contains approximately 85 mg of caffeine).
* Subject plans consumption of alcohol, or consumption of caffeine within 48 hours of study conduct or throughout the entire dosing and evaluation period of the study.
* (Females only): Subject is pregnant or lactating.
* Subject has participated in another investigational drug, medical device, or biologics study within 30 days prior to dosing.

formed on all females).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Vasoconstriction response | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Lehman,, M.Sc., Principal Investigator — DermTech International
Locations (1):
- DermTech International, San Diego, California, United States